CLINICAL TRIAL: NCT02501265
Title: Randomized Controlled Smoking Cessation Trial on Adaptive Pharmacotherapy
Brief Title: Adaptive Pharmacotherapy for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00072077; P50DA027840 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-17 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Bupropion; Varenicline; Adaptive Approach; Nicotine Patch; Chantix
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: The study (N=300) is a double-blinded randomized placebo-controlled trial designed to compare biochemically-confirmed abstinence rates in smokers randomized to Varenicline Adaptive Protocol vs. Varenicline (N=150) and for comparison, Nicotine Patch Adaptive Protocol vs. Nicotine Patch (N=150).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Varenicline Standard Protocol (Active Comparator): Participant choses Varenicline-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Varenicline. Consistent with Varenicline Standard Treatment, 1 week prior to the TQD the participant will switch to active Varenicline and placebo Bupropion. Participant will continue active Varenicline and placebo Bupropion to 12 weeks post-TQD.
  Interventions: Behavioral: Varenicline Standard Protocol
- Nicotine Patch Standard Protocol (Active Comparator): Participant choses Nicotine patch-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Nicotine Patch. One week prior to TQD, participant will start placebo Bupropion. Consistent with Nicotine Patch Standard Treatment, participant will start active Nicotine Patch on TQD. Participant will continue active Nicotine Patch and placebo Bupropion to 12 weeks post-TQD.
  Interventions: Behavioral: Nicotine Patch Standard Protocol
- Varenicline Adaptive Protocol (Experimental): Participant chooses Varenicline treatment and is randomized to Adaptive Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts active Varenicline. Two weeks prior to TQD, cigarettes smoked per day is assessed. If the number of cigarettes smoked per day is reduced by >50%, the participant is considered a Varenicline responder, and starts placebo Bupropion 1 week prior to the TQD. If the participant DOES NOT reduce cigarettes smoked per day by >50%, the participant is considered a Varenicline non-responder and starts active Bupropion 1 week prior to TQD. Varenicline responders will continue active Varenicline and placebo Bupropion to 12 weeks post TQD. Varenicline non-responders will continue active Varenicline and active Bupropion to 12 weeks post TQD.
  Interventions: Drug: Varenicline Adaptive Protocol
- Nicotine Patch Adaptive Protocol (Experimental): Participant choses Nicotine treatment and is randomized to Adaptive Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts active Nicotine Patches. Two weeks prior to TQD, cigarettes smoked per day is assessed. If cigarettes smoked per day is reduced by >50%, the participant is considered a Nicotine Patch responder and starts placebo Bupropion 1 week prior to the TQD. If the participant DOES NOT reduce cigarettes smoked per day by >50%, the participant is considered a Nicotine Patch non-responder and starts active Bupropion 1 week prior to the TQD. Nicotine Patch responders will continue active Nicotine Patches and placebo Bupropion to 12 weeks post TQD. Nicotine Patch non-responders will continue active Nicotine Patches and Bupropion to 12 weeks post TQD.
  Interventions: Drug: Nicotine Adaptive Protocol

INTERVENTIONS:
Behavioral: Varenicline Standard Protocol — 4 weeks pre-TQD: Start Placebo Varenicline
  1 week prior to TQD: Switch to Active Varenicline
  1 week prior to TQD: Start Placebo Bupropion Varenicline + Placebo Bupropion to 12 weeks post TQD
  Other Names: Standard Varenicline
  Arms: Varenicline Standard Protocol
Behavioral: Nicotine Patch Standard Protocol — 4 weeks pre-TQD: Start Placebo Nicotine Patch TQD: Start active Nicotine Patch
  1 week prior to TQD: Start Placebo Bupropion Nicotine Patch + Placebo Bupropion to 12 weeks post TQD
  Other Names: Standard Nicotine Patch
  Arms: Nicotine Patch Standard Protocol
Drug: Varenicline Adaptive Protocol — VARENICLINE RESPONDER 4 weeks pre-TQD: Start Varenicline 2 weeks pre-TQD: DOES reduce cigs/day by > 50% 1 week pre-TQD: Start Placebo Bupropion Varenicline + Placebo Bupropion to 12 weeks post TQD
  VARENICLINE NON-RESPONDER 4 weeks pre-TQD: Start Varenicline 2 weeks pre-TQD: DOES NOT reduce cigs/day by > 50%
  1 week pre-TQD: Start active Bupropion Varenicline + Bupropion to 12 weeks post TQD
  Other Names: Adaptive Varenicline
  Arms: Varenicline Adaptive Protocol
Drug: Nicotine Adaptive Protocol — NICOTINE PATCH RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES reduce cigs/day by > 50% 1 week pre-TQD: Start Placebo Bupropion Patch + Placebo Bupropion to 12 weeks post TQD
  NICOTINE PATCH NON-RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES NOT reduce cigs/day by > 50%
  1 week pre-TQD: Start Bupropion Patch + Bupropion to 12 weeks post TQD
  Other Names: Adaptive Nicotine
  Arms: Nicotine Patch Adaptive Protocol

SUMMARY:
The purpose of this study is to assess an "adaptive" approach to smoking cessation pharmacotherapy. The protocol is designed to compare adaptive vs. standard approaches to two common smoking cessation pharmacotherapies - Varenicline (commonly known as Chantix) and the Nicotine Patch. The investigators hypothesize that participants allocated to adaptive therapy will show significantly higher biochemically confirmed 30-day continuous abstinence at 12 weeks post-Target Quit Day (TQD).

DETAILED DESCRIPTION:
The purpose of this study is to assess an "adaptive" approach to smoking cessation pharmacotherapy. The protocol is designed to compare adaptive vs. standard approaches to two common smoking cessation pharmacotherapies (Varenicline and Nicotine Patch). The adaptive treatment approach provides the addition of Bupropion in the pre-quit period for participants who are not "responding" to initial treatment. Little is known about the adaptive use of Varenicline or Nicotine Patch, in which Bupropion is added to Varenicline or Patch for those who do not respond to one of these medications in a pre-quit treatment period. This study attempts to address these knowledge deficits. The study (N=300) is a double-blinded randomized placebo-controlled trial designed to compare biochemically-confirmed abstinence rates in smokers randomized to Varenicline Adaptive Protocol vs. Varenicline (N=150) and for comparison, Nicotine Patch Adaptive Protocol vs. Nicotine Patch (N=150). The "Varenicline Adaptive Protocol" is conducted by starting treatment with Varenicline 4 weeks prior to the quit day and following each participant's response to this pre-treatment medication. After 2 weeks, if the patient shows a reduction greater than 50% in cigarettes smoked per day, then the patient is considered to be a "Varenicline responder" and is continued on Varenicline alone out to 12-weeks post quit day. If the patient does not spontaneously decrease smoking in the pre-quit period by more than 50% cigarettes per day, the patient is considered to be a "Varenicline non-responder" and Bupropion is added to the Varenicline. For comparison, an identical protocol is used with nicotine patch vs. nicotine patch adaptive treatment. The study uses only FDA-approved medications: Varenicline, Nicotine Patch, Bupropion, and placebo controls. To pattern clinical practice, participants will be able to choose whether they would like to use a patch or Varenicline-based treatment. After choosing, however, they will be randomized to adaptive vs. non-adaptive version of that treatment. Placebo medications are matched throughout the study. Participants will be blinded to all medications. All participants will receive behavioral treatment including a single 40-minute visit with a medical provider. The study is designed to provide researchers and clinicians with a better understanding of how to use adaptive pharmacotherapy protocols to improve smoking cessation rates.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older
2. Actively smoking 5 or more cigarettes per day for at least one year
3. Fluency in spoken and written English
4. Willing to set a quit date within 6 weeks
5. Access to a telephone
6. Willingness to take Varenicline OR nicotine patch (patient choice)
7. Willingness to take Bupropion

Exclusion Criteria

1. Daily use of a second form of tobacco or nicotine (e.g. e-cigarettes, cigars, chewing tobacco, snuff).
2. Current use of a smoking cessation medication (e.g. nicotine replacement, Varenicline, Bupropion).
3. Report of pregnancy, attempting to get pregnant, or actively breast feeding or positive urine pregnancy test (only given to females with child bearing potential).
4. Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, M.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis JM, Masclans L, Rose JE. Adaptive Smoking Cessation Using Precessation Varenicline or Nicotine Patch: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332214. doi: 10.1001/jamanetworkopen.2023.32214. PMID 37682573

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline Standard Protocol: Participant chooses Varenicline-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Varenicline. Consistent with Varenicline Standard Treatment, 1 week prior to the TQD the participant will switch to active Varenicline and placebo Bupropion. Participant will continue active Varenicline and placebo Bupropion to 12 weeks post-TQD.
  Varenicline Standard Protocol: 4 weeks pre-TQD: Start Placebo Varenicline 1 week prior to TQD: Switch to Active Varenicline
  1 week prior to TQD: Start Placebo Bupropion Varenicline + Placebo Bupropion to 12 weeks post TQD
- Nicotine Patch Standard Protocol: Participant chooses Nicotine patch-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Nicotine Patch. One week prior to TQD, participant will start placebo Bupropion. Consistent with Nicotine Patch Standard Treatment, participant will start active Nicotine Patch on TQD. Participant will continue active Nicotine Patch and placebo Bupropion to 12 weeks post-TQD.
  Nicotine Patch Standard Protocol: 4 weeks pre-TQD: Start Placebo Nicotine Patch TQD: Start active Nicotine Patch
  1 week prior to TQD: Start Placebo Bupropion Nicotine Patch + Placebo Bupropion to 12 weeks post TQD
- Varenicline Adaptive Protocol: Participant chooses Varenicline treatment and is randomized to Adaptive Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts active Varenicline. Two weeks prior to TQD, cigarettes smoked per day is assessed. If the number of cigarettes smoked per day is reduced by >50%, the participant is considered a Varenicline responder, and starts placebo Bupropion 1 week prior to the TQD. If the participant DOES NOT reduce cigarettes smoked per day by >50%, the participant is considered a Varenicline non-responder and starts active Bupropion 1 week prior to TQD. Varenicline responders will continue active Varenicline and placebo Bupropion to 12 weeks post TQD. Varenicline non-responders will continue active Varenicline and active Bupropion to 12 weeks post TQD.
  Varenicline Adaptive Protocol: VARENICLINE RESPONDER 4 weeks pre-TQD: Start Varenicline 2 weeks pre-TQD: DOES reduce cigs/day by > 50% 1 week pre-TQD: Start Placebo Bupropion Varenicline + Placebo Bupropion to 12 weeks post TQD
  VARENICLINE NON-RESPONDER 4 weeks pre-TQD: Start Varenicline 2 weeks pre-TQD: DOES NOT reduce cigs/day by > 50%
  1 week pre-TQD: Start active Bupropion Varenicline + Bupropion to 12 weeks post TQD
- Nicotine Patch Adaptive Protocol: Participant chooses Nicotine treatment and is randomized to Adaptive Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts active Nicotine Patches. Two weeks prior to TQD, cigarettes smoked per day is assessed. If cigarettes smoked per day is reduced by >50%, the participant is considered a Nicotine Patch responder and starts placebo Bupropion 1 week prior to the TQD. If the participant DOES NOT reduce cigarettes smoked per day by >50%, the participant is considered a Nicotine Patch non-responder and starts active Bupropion 1 week prior to the TQD. Nicotine Patch responders will continue active Nicotine Patches and placebo Bupropion to 12 weeks post TQD. Nicotine Patch non-responders will continue active Nicotine Patches and Bupropion to 12 weeks post TQD.
  Nicotine Adaptive Protocol: NICOTINE PATCH RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES reduce cigs/day by > 50% 1 week pre-TQD: Start Placebo Bupropion Patch + Placebo Bupropion to 12 weeks post TQD
  NICOTINE PATCH NON-RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES NOT reduce cigs/day by > 50%
  1 week pre-TQD: Start Bupropion Patch + Bupropion to 12 weeks post TQD
Period: Overall Study
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Started | 63 | 30 | 64 | 31
Completed | 46 | 21 | 46 | 23
Not Completed | 17 | 9 | 18 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol | Total
Number analyzed (Participants) | 63 | 30 | 64 | 31 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.5) | 45.0 (16.3) | 49.1 (12.6) | 50.3 (11.6) | 49.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 35 | 19 | 101
  Male | 33 | 13 | 29 | 12 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 62 | 30 | 63 | 29 | 184
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 23 | 21 | 19 | 17 | 80
  White | 38 | 6 | 41 | 13 | 98
  More than one race | 1 | 2 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-confirmed 30-day Continuous Smoking Abstinence
Description: Number of participants who self report complete smoking abstinence over the last 30 days and are also verified to be abstinent by carbon monoxide (CO) expired breath testing with CO < 7 parts per million.
Time Frame: 12 weeks post-TQD (Visit 4)
Population: Intent-to-treat analysis of a clinical population with significant comorbidity and minimal exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Number analyzed (Participants) | 63 | 30 | 64 | 31
Participants | 5 | 3 | 18 | 5

2. Secondary Outcome: 7-day Point Prevalence Biochemically Confirmed Abstinence
Description: Number of participants who self report complete smoking abstinence over the last 7 days and are also verified to be abstinent by carbon monoxide (CO) expired breath testing with CO < 7 parts per million.
Time Frame: 12 weeks post-TQD (Visit 4)
Population: Intent-to-treat analysis of a clinical population with significant comorbidity and minimal exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Number analyzed (Participants) | 63 | 30 | 64 | 31
Participants | 6 | 3 | 23 | 6

3. Secondary Outcome: Phone-assessed Self-reported Abstinence
Description: Number of participants who self reported smoking abstinence over the last 24 hours assessed via single-item question.
Time Frame: 52 weeks post-TQD
Population: Intent-to-treat analysis of a clinical population with significant comorbidity and minimal exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Number analyzed (Participants) | 63 | 30 | 64 | 31
Participants | 16 | 5 | 21 | 6

4. Secondary Outcome: Change in Cigarettes Smoked Per Day
Description: The percentage of participants who decreased the number of daily cigarettes smoked by 50% or more from the baseline assessment visit to 12 weeks post target quit day assessment visit collected by self-report in participants who completed the 12-week post target quit day assessment visit
Time Frame: 12 weeks post-TQD (Visit 4)
Population: Analysis of a clinical population with significant comorbidity and minimal exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Number analyzed (Participants) | 56 | 25 | 59 | 28
percentage of participants | 80.4 | 71.4 | 89.4 | 82.6

5. Secondary Outcome: Change in Cigarettes Smoked Per Day (Phone)
Description: The percentage of participants who decreased the number of daily cigarettes smoked by 50% or more from the baseline assessment visit to 52 weeks post target quit day assessment visit collected by self-report in participants who completed the 52-week post target quit day phone assessment.
Time Frame: 52 weeks post-TQD
Population: Analysis of a clinical population with significant comorbidity and minimal exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
Number analyzed (Participants) | 51 | 24 | 54 | 28
percentage of participants | 67.6 | 57.1 | 84.8 | 62.5

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were collected in such a manner that specific adverse event terms cannot be separated or categorized. Specifically, participants were provided with open ended questions at each study visit to assess any symptom that might have occurred, and were asked to provide a description of these symptoms in their own words. What is reported below is total percentage of participants who reported adverse events of any kind.
Groups:
- Varenicline Standard Protocol: Participant choses Varenicline-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Varenicline. Consistent with Varenicline Standard Treatment, 1 week prior to the TQD the participant will switch to active Varenicline and placebo Bupropion. Participant will continue active Varenicline and placebo Bupropion to 12 weeks post-TQD.
  Varenicline Standard Protocol: 4 weeks pre-TQD: Start Placebo Varenicline 1 week prior to TQD: Switch to Active Varenicline
  1 week prior to TQD: Start Placebo Bupropion Varenicline + Placebo Bupropion to 12 weeks post TQD
- Nicotine Patch Standard Protocol: Participant choses Nicotine patch-based treatment and is then randomized to Standard Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts placebo Nicotine Patch. One week prior to TQD, participant will start placebo Bupropion. Consistent with Nicotine Patch Standard Treatment, participant will start active Nicotine Patch on TQD. Participant will continue active Nicotine Patch and placebo Bupropion to 12 weeks post-TQD.
  Nicotine Patch Standard Protocol: 4 weeks pre-TQD: Start Placebo Nicotine Patch TQD: Start active Nicotine Patch
  1 week prior to TQD: Start Placebo Bupropion Nicotine Patch + Placebo Bupropion to 12 weeks post TQD
- Nicotine Patch Adaptive Protocol: Participant choses Nicotine treatment and is randomized to Adaptive Treatment arm (N=75). Four weeks prior to target quit date (TQD), participant starts active Nicotine Patches. Two weeks prior to TQD, cigarettes smoked per day is assessed. If cigarettes smoked per day is reduced by >50%, the participant is considered a Nicotine Patch responder and starts placebo Bupropion 1 week prior to the TQD. If the participant DOES NOT reduce cigarettes smoked per day by >50%, the participant is considered a Nicotine Patch non-responder and starts active Bupropion 1 week prior to the TQD. Nicotine Patch responders will continue active Nicotine Patches and placebo Bupropion to 12 weeks post TQD. Nicotine Patch non-responders will continue active Nicotine Patches and Bupropion to 12 weeks post TQD.
  Nicotine Adaptive Protocol: NICOTINE PATCH RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES reduce cigs/day by > 50% 1 week pre-TQD: Start Placebo Bupropion Patch + Placebo Bupropion to 12 weeks post TQD
  NICOTINE PATCH NON-RESPONDER 4 weeks pre-TQD: Start Patch 2 weeks pre-TQD: DOES NOT reduce cigs/day by > 50%
  1 week pre-TQD: Start Bupropion Patch + Bupropion to 12 weeks post TQD
Arm/Group | Varenicline Standard Protocol | Nicotine Patch Standard Protocol | Varenicline Adaptive Protocol | Nicotine Patch Adaptive Protocol
All-Cause Mortality (participants affected / at risk) | 1/63 | 0/30 | 0/64 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/30 | 1/64 | 0/31
Other Adverse Events (participants affected / at risk) | 48/63 | 25/30 | 58/64 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Standard Protocol (N=63) | Nicotine Patch Standard Protocol (N=30) | Varenicline Adaptive Protocol (N=64) | Nicotine Patch Adaptive Protocol (N=31)
Hospitalization related to pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Standard Protocol (N=63) | Nicotine Patch Standard Protocol (N=30) | Varenicline Adaptive Protocol (N=64) | Nicotine Patch Adaptive Protocol (N=31)
Report of any: Vivid Dreams, Constipation, Dry Mouth, Dizziness, Headache, Insomnia, Nausea, Anxiety (General disorders) | 48 (48) | 25 (25) | 58 (58) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02501265/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT02501265/ICF_001.pdf